CLINICAL TRIAL: NCT00640523
Title: Phase II Study of Forodesine in Subjects With Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCX1777-210
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: forodesine HCl — 2 x 100mg capsules daily

SUMMARY:
To evaluate the effectiveness and safety of forodesine in CLL patients

DETAILED DESCRIPTION:
To investigate the efficacy (complete response [CR] + partial response [PR]) of forodesine in treating subjects with CLL who have failed at least one prior treatment regimen or who are treatment naïve but are either elderly, have poor performance status or are otherwise predicted not to tolerate cytotoxic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. Diagnosis of CLL established by peripheral blood and/or bone marrow examination and using the standard diagnostic criteria.
3. Subjects with Rai stage III or IV, or earlier stage requiring therapy as determined by the 1996 National Cancer Institute -Working Group (NCI-WG) criterion
4. Primary resistant (no CR or PR) or progressive disease after response to at least one prior treatment regimen OR treatment naïve subjects who meet at least one of the following criteria.

   1. age >65 years
   2. Eastern Cooperative Oncology Group (ECOG) performance status of 2, 3, or 4
   3. Inability to tolerate standard cytotoxic chemotherapy in the opinion of the treating physician.
5. ECOG performance status of 0, 1, or 2 (for subjects with primary resistance or progressive disease after response to at least one prior treatment regimen).
6. Willing to take adequate contraceptive measures (i.e., latex condom, cervical cap, diaphragm, abstinence, etc.) for the entire duration of the study and 3 months after, except for patients who are post menopausal or have prior hysterectomy.
7. All investigational treatments should have been discontinued for at least 3 weeks prior to the initiation of the study drug.

Exclusion Criteria:

1. Pregnant or nursing.
2. Unable or unwilling to sign consent.
3. Severe, ongoing co-morbid conditions, which would preclude safe delivery of the investigational therapy.
4. Active serious infections that are not controlled by antibiotics.
5. ECOG performance status >2 (except for treatment naïve subjects where ECOG performance status 0, 1 or 5 is excluded).
6. Inadequate renal function: creatinine > or equal to 2.0 unless related to the disease.
7. Inadequate liver function: bilirubin > or equal to 3.0; transaminases > or equal to 3.0 times the upper limit of normal unless related to the disease.
8. Known positive test for human immunodeficiency virus (HIV).
9. Subjects with known hepatitis B and/or hepatitis C active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-03; Primary Completion 2010-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Up to 6 cycles of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Asher Chanan-Khan, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (11):
- United States (8):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - UCLA Medical Center, Los Angeles, California
  - Indiana University Cancer Pavillion, Indianapolis, Indiana
  - Center for Cancer & Blood Disorders, PC, Bethesda, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medical College, New York, New York
  - Oregon Health & Science University, Portland, Oregon
- Australia (3):
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Frankston Hospital, Frankston, Victoria
  - Cabrini Hospital, Malvern, Victoria